CLINICAL TRIAL: NCT04317456
Title: AChild - Austrian Children With Hearing Impairment - Longitudinal Database
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: AChild
Record Dates: First submitted 2020-02-27; First posted 2020-03-23 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hearing Impaired Children
Keywords: Longitudinal Database
MeSH Terms: interventions — Hearing Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hearing Aids and Hearing Implants — Hearing Aids and Hearing Implants (age at first fitting and implantation and aided audibility)
Behavioral: Family Centred Early Intervention — Family Centred Early Intervention

SUMMARY:
There is high variability in outcomes in children with hearing impairment. Existing literature focus mainly on subpopulations (children with hearing aids, children with CI) and is usually not epidemiological. Often children with additional needs (intellectual disability, visual impairment, autism spectrum disorder, complex syndromes) are excluded from the studies. This subgroup of children makes up around 1/3 of the population of children with hearing impairment.

What factors contribute to the unexplained variance in language development in children with hearing loss? (including children with additional needs, multilingual) There is a lack of European epidemiological studies that evaluate the effects of Newborn Hearing Screening and early intervention.

DETAILED DESCRIPTION:
Aims:

* to collect population based data on children born in Upper Austria with a significant hearing impairment and to describe this population in detail regarding audiological, etiological (including geno- and phenotypical correlations), neurodevelopmentally, psychological, psychiatrically and linguistically with a special interest is in children with additional needs
* collecting child development outcomes (language, communication, psychosocial) and family outcomes (quality of life, stress)
* to investigate possible effects of the Newborn Hearing Screening, early intervention and specific parent behaviors targeted in early intervention
* collecting developmental trajectories of the total sample and subgroups of the sample (particularly audiological, etiological and cognitive). This data should help identify red flags
* investigating predictors of developmental trajectories regarding the child and the intervention (e.g. time and

Hypothesis:

* It is expected that .2% of the total population of preschool children have a sensorineural hearing loss (bilateral and unilateral)
* a significantly higher prevalence of intellectual disabilities (up to 20%), visual impairment, autism spectrum disorder and motor impairment
* it is expected that for at least 50% of the children, there is a genetic explanation for the hearing impairment and 30% out of them are expected to be syndromal
* it is expected that there is a higher proportion of children with psycho-social problems (especially peer problems and behavioral-/emotional problems)
* Due to a change in the environmental conditions over the past two decades, better child outcomes, compared to previous ones are expected. Nevertheless around 30-50% of the children are expected to not be reaching their nonverbal cognitive potential.
* expected intervention effects, particularly for provision with and use of hearing technology family-child interaction self-efficacy and wellbeing of the family regulated media use

ELIGIBILITY:
Inclusion Criteria:

* with significant sensorineural hearing impairment or permanent congenital conductive deafness; profound hearing impairment above frequency of 0.5, 1, 2 and 4 kHz of ≥ 25 dB
* unilateral or bilateral
* diagnosed before the age of 6 years
* including children with multiple disabilities
* including children with another language than German (including sign language)
* including children with auditory neuropathy spectrum disorder (ANS)
* including children with behavioral problems and psychiatric disorders

Exclusion Criteria:

* children who were older than 6 years when they were diagnosed
* who's families do not agree to participate in the study
* with temporary conductive deafness

Max Age: 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children in Upper Austria with a significant sensorineural hearing impairment or permanent congential conductive deafness who were diagnosed before the age of 6 years are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Vocabulary Expressive of the Child | 5 years
  Questionnaire used for this Outcome is:
  SET 3-5
Vocabulary Receptive of the Child | 5 years
  Questionnaire used for this Outcome is:
  PPVT-4
Grammar Expressive of the Child | 5 years
  Questionnaire used for this Outcome is:
  LOGIK_S Expressive Grammatik
Language Receptive of the Child | 5 years
  Questionnaire used for this Outcome is:
  TROG-D
Language Receptive of the Child (ÖGS) | 5 years
  Questionnaire used for this Outcome is:
  RDLS ÖGS
Social Communication of the Child | 5 years
  Questionnaire used for this Outcome is:
  CCC-2
Symbolic Behaviour of the Child | 5 years
  Questionnaire used for this Outcomes is:
  CSBS
Psychosocial Development of the Child | 5 years
  Questionnaire used for this Outcome is:
  SDQ
Emotional and Behaviour Problems of the Child | 5 years
  Questionnaire used for this Outcome is:
  CBCL
Quality of Life of the Child | 5 years
  Questionnaire used for this Outcome is:
  AUQUEI
Family Stress | 5 years
  Questionnaire used for this Outcome is:
  EBI (Elternbelastungsinventar)
Parental Self-Efficacy | 5 years
  Questionnaire used for this Outcome is:
  SPISE-R
Non-Verbal Development | 5 years
  Questionnaire used for this Outcome is:
  SON

SECONDARY OUTCOMES:
Executive Functioning of the Child | 5 years
  The questionnaire used for this Outcome is:
  VIEF (Verhaltens - Inventar Exekutiver Funktionen)
Adaptive Skills of the Child | 5 years
  The questionnaire used for this Outcome is:
  Vineland-2
Visual successive memory and attention | 5 years
  The questionnaire used for this Outcome is:
  KNOX cube test
Phonological working memory | 5 years
  The questionnaire used for this Outcome is:
  Mottier test
Mental Health | 5 years
  The questionnaire used for this Outcome is:
  SDQ 4-16 (Strength and Difficulties Questionnaire)
Media use | 5 years
  The questionnaire used for this Outcome is:
  Kinder und Medien Fragebogen

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Kepler University, Linz, Austria

IPD SHARING:
Plan to Share IPD: Undecided